CLINICAL TRIAL: NCT05607420
Title: Open-label Dose-finding and Dose-expansion Study to Evaluate the Safety, Expansion, Persistence, and Clinical Activity of UCART20x22 in Subjects With Relapsed or Refractory B-Cell Non-Hodgkin Lymphoma (B-NHL)
Brief Title: Study Evaluating UCART20x22 in B-Cell Non-Hodgkin Lymphoma
Acronym: NatHaLi-01
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cellectis S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCART20x22_01
Record Dates: First submitted 2022-10-25; First posted 2022-11-07 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: B-cell Non-Hodgkin Lymphoma (B-NHL)
Keywords: B-cell Non-Hodgkin Lymphoma (B-NHL); Relapsed/Refractory B-NHL; Universal Chimeric Antigen Receptor T-Cell (UCAR-T) Therapy; Allogeneic; Transcription Activator-Like Effector Nuclease (TALEN®)
MeSH Terms: conditions — Lymphoma, B-Cell; Recurrence | interventions — Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose finding part (Experimental): UCART20x22 tested at several dose levels until the Maximum Tolerated Dose (MTD) and/or the Recommended Phase 2 Dose (RP2D) is identified.
  Dose expansion part: UCART20x22 administered at the RP2D determined during the dose finding part
  Interventions: Biological: UCART20x22; Biological: CLLS52

INTERVENTIONS:
Biological: UCART20x22 — Allogeneic engineered T-cells expressing anti-CD20 and anti-CD22 Chimeric Antigen Receptors given following a lymphodepletion regimen
Biological: CLLS52 — A monoclonal antibody that recognizes a CD52 antigen
  Other Names: Alemtuzumab

SUMMARY:
First-in-human, open-label, dose-finding and dose-expansion study of UCART20x22 administered intravenously in subjects with relapsed or refractory B-Cell Non-Hodgkin Lymphoma (B-NHL). The purpose of this study is to evaluate the safety and clinical activity of UCART20x22 and determine the Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D).

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Relapsed or refractory (R/R) mature B-NHL per 2016 WHO criteria and positive for CD20 and/or CD22
* Subjects with NHL subtypes defined by WHO:
* Dose-Finding Part: R/R mature B-NHL (except chronic lymphocytic leukemia/small lymphocytic leukemia [CLL/SLL], Richter's transformation from prior CLL/SLL, Burkitt's lymphoma, and Waldenstrom's macroglobulinemia)
* Dose-Expansion Part: R/R LBCL, defined as:

  i. DLBCL; ii. High-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements; iii. Transformed FL or transformed marginal zone lymphoma (MZL); iv. Follicular lymphoma Grade 3B
* R/R disease after at least 2 lines of prior treatment, which must have included:
* An Anti-CD20 MoAb and an anthracycline for DLBCL, high-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements, primary mediastinal large B-cell lymphoma (PMBCL), or transformed FL or MZL
* An alkylating agent in combination with an anti-CD20 MoAb for FL
* An anthracycline or bendamustine-containing chemotherapy regimen and a Bruton's tyrosine kinase (BTK) inhibitor for mantle cell lymphoma (MCL)
* Autologous anti-CD19 CAR T-cell therapy, if approved and available for the indicated lymphoma subtype, unless the subject is unable or is ineligible to receive approved autologous anti-CD19 CAR T-cell therapy (e.g., fail leukapheresis or manufacture, unable to wait for manufacture, CD19 negative disease, etc.)
* Autologous hematopoietic stem cells must be available prior to the start of the LD regimen if the subject is considered high-risk for prolonged hematologic toxicity.

Exclusion Criteria:

* Prior use of an investigational product (except for cell or gene therapies and MoAbs) within 5 half-lives or within 14 days, whichever is shorter, prior to start of LD regimen
* Previous approved therapy including chemotherapy, biologic (except MoAbs), or targeted therapy for R/R B-NHL with 5 half-lives or within 14 days, whichever is shorter, prior to start of the LD regimen
* > 4 lines of therapy R/R B-NHL prior to start of the LD regimen.
* Prior MoAb therapy (approved or investigational) within 30 days prior to start of LD
* Prior systemic immunostimulatory agent within 3 half-lives prior to start of the LD regimen
* Prior cell or gene therapy (approved or investigational) within 6 months of the start of LD
* Prior cell or gene therapy (approved or investigational) targeting both CD20 and CD22
* Autologous HSCT infusion within 6 weeks of the start of LD
* Allogeneic HSCT within 3 months of the start of LD, or donor lymphocyte infusion within 6 weeks of the start of LD
* Active acute or chronic graft versus host disease (GvHD). Subjects should be off all immunosuppressive therapies for at least 6 weeks prior to start of LD
* Radiotherapy within 8 weeks (except for palliative radiotherapy for specific on-target lesions) (prior to start of LD regimen)
* Evidence of active central nervous system (CNS) lymphoma or previous CNS involvement of R/R B-NHL
* Presence of an active and clinically relevant CNS disorder
* Daily treatment with >20 mg prednisone or equivalent
* Known active infection, or reactivation of a latent infection, whether bacterial or viral, fungal, mycobacterial, or other pathogens
* History of hypersensitivity to alemtuzumab
* History of neutralizing anti-drug antibody against alemtuzumab
* Any known uncontrolled cardiovascular disease within 3 months of enrollment
* Subjects requiring immunosuppressive treatment
* Major surgery within 28 days prior to start of LD
* Evidence of another uncontrolled malignancy within 2 years prior to Screening (except in situ nonmelanoma skin cell cancers and/or carcinoma in-situ of the cervix)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Dose finding and expansion parts: Incidence of adverse events/serious adverse events/dose limiting toxicity [Safety and Tolerability] | From study entry through month 12
  Incidence, nature and severity of adverse events and serious adverse events in relation to UCART20x22 and/or lymphodepletion
Dose finding part: Occurrence of Dose Limiting Toxicities (DLTs) | Up to Day 28 post UCART20x22 infusion

SECONDARY OUTCOMES:
Investigator assessed overall response rate (ORR) according to Lugano Response Criteria for Malignant Lymphoma | At Day 28, Day 84, Month 6, Month 9, Month 12
Duration of Response | From achievement of the initial response to disease relapse/progression or death from any cause, assessed up to Month 12
Progression-free survival (PFS) | From the first day of any study treatment to the date of disease progression or death from any cause, whichever occurs first, assessed up to Month 12
Overall survival | From initiation of any study treatment to death from any cause, assessed up to Year 15

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Abramson, MD, Principal Investigator — Harvard Medical School - Massachusetts General
Locations (10):
- United States (4):
  - The University of Chicago Medical Center (UCMC), Chicago, Illinois
  - Harvard Medical School - Massachusetts General Hospital, Boston, Massachusetts
  - Rutgers Cancer Institute of New Jersey (CINJ) - New Brunswick, New Brunswick, New Jersey
  - Sarah Cannon - St. David South Austin Medical Center, Austin, Texas
- France (4):
  - Hospices Civils de Lyon (HCL) - Centre Hospitalier Lyon-Sud, Pierre-Bénite, Auvergne Rhone Alpe
  - Centre Hospitalier Universitaire de Montpellier (CHU Montpellier) - Hopital Saint-Eloi, Montpellier, Occitanie
  - Centre Hospitalier Universitaire de Nantes (CHU de Nantes)-Hotel-Dieu, Nantes
  - Assistance Publique-Hopitaux de Paris (AP-HP) - Hopital Saint-Louis - Centre Integre en Cancerologie, Paris, Île-de-France Region
- Spain (2):
  - Universidad de Navarra - Clinica Universidad de Navarra (CUN) - Pamplona, Pamplona, Navarre
  - Hospital Universitario Virgen del Rocio (HUVR) - Instituto de Biomedicina de Sevilla (IBIS), Seville

IPD SHARING:
Plan to Share IPD: No